CLINICAL TRIAL: NCT05606783
Title: Using Bluetooth Home Blood Pressure Monitors With Pharmacist Interventions to Manage Uncontrolled Hypertension in the Community Setting - A Pilot Study
Brief Title: Using Bluetooth Home Blood Pressure Monitors With Pharmacist Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: National Association of Chain Drug Stores (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00036888
Record Dates: First submitted 2019-03-26; First posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2019-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Surveys and Questionnaires; Equipment and Supplies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Home blood pressure monitoring (Experimental): * Smart Phones with Apple Health Software will be used to monitor blood pressure once a day, and results will be sent automatically to the patients EHR (Epic)
  * The Omron 10 Series Wireless Upper Arm Blood Pressure Device will be given to the patient to monitor blood pressure at home daily
  * Patients will be scheduled for a one-hour in-person appointment for the initial study visit where informed consent will be obtained, and for the final study visit
  Interventions: Behavioral: Telehealth Follow-up Visits; Behavioral: Surveys; Device: Devices

INTERVENTIONS:
Behavioral: Telehealth Follow-up Visits — • Follow-up with patients once per week for six (6) weeks via scheduled 20-minute telehealth appointment with each patient via the HIPAA secure and compliant platform, VSee
  o During this telehealth appointment, the study pharmacists will counsel the patients on their blood pressure readings for that week and provide lifestyle education focusing on patient-specific diet and exercise recommendations
Behavioral: Surveys — A pre- and post-survey will be given at the initial and final in-person appointments, respectively
  • These surveys will collect basic patient demographics, knowledge of blood pressure, comfort with checking blood pressure at home, and previous experience working with a pharmacist
Device: Devices — Smart Phones with Apple Health Software will be used to monitor blood pressure once a day, and results will be sent automatically to the patients EHR (Epic)
  • The Omron 10 Series Wireless Upper Arm Blood Pressure Device will be given to the patient to monitor blood pressure at home daily

SUMMARY:
Family Medicine patients with uncontrolled hypertension will be given a Bluetooth enabled home blood pressure machine to monitor their blood pressure every day for 6 weeks. The blood pressure results will be sent automatically to the patient's electronic medical record via applications on their iPhone. Study pharmacists will follow-up with the patients once per week via a telehealth appointment using the app VSee, where the blood pressure results will be reviewed. The pharmacists will also counsel the patients on lifestyle modifications in order to improve blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* must be at least 18 years old
* have a smartphone compatible with the mobile intervention (iPhone)
* have been previously diagnosed with hypertension
* have uncontrolled hypertension (SBP > 130 mmHg and/or DBP > 80 mmHg)
* be under the care of a primary care physician in the Family Medicine Department of the USF Morsani Center for Advanced Care
* have had at least one prescription filled at Pharmacy Plus within the last six months
* speaks English fluently

Exclusion Criteria:

* already under the care of a clinical pharmacist in the Family Medicine department
* pregnant
* have a serious existing medical condition(s) that may affect their ability to self-monitor their blood pressure (for example, stroke, dementia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Comfort | 8 weeks
  Patient comfort in using home telemonitoring for blood pressure combined with pharmacist counseling and monitoring will be measured using a survey instrument with a Likert scale (4-point scale). (Most of the time; Some of the time; Seldom; Never) (Strongly agree; Agree; Disagree; Strongly disagree) (Nothing; Very little; Some; Knowledgeable)

SECONDARY OUTCOMES:
Determine if pharmacists' interventions improved BP | 8 weeks
  BP readings were reported and evaluated to discover if these were improved with pharmacists' interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy H Updike, PharmD, Principal Investigator — University of South Florida College of Pharmacy
Locations (1):
- USF Pharmacy Plus, Tampa, Florida, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/83/NCT05606783/Prot_SAP_000.pdf
  • Informed Consent Form (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/83/NCT05606783/ICF_001.pdf